CLINICAL TRIAL: NCT05750264
Title: Efficacy of Intravenous Ibuprofen in Multimodal Pain Management After Open Abdominal Hysterectomy: A Randomised Trial
Brief Title: Intravenous Ibuprofen Postoperative Analgesia After Abdominal Hysterectomy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Abd-Elazeem Abd-Elhameed Elbakry, Professor, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2/2023 ANET10-1
Record Dates: First submitted 2023-02-12; First posted 2023-03-01 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Post Operative Analgesia
MeSH Terms: interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ibuprofen group (Active Comparator): intravenous ibuprofen 800mg in 200 ml normal saline+IV paracetamol 1000mg+Transversus abdominis plane block
  Interventions: Drug: Ibuprofen
- Control group (No Intervention): 200 ml normal saline+IV paracetamol1000mg+Transversus abdominis plane block

INTERVENTIONS:
Drug: Ibuprofen — 800 mg of IV ibuprofen
  Arms: ibuprofen group

SUMMARY:
The current research is designed to investigate the analgesic efficacy of intravenous ibuprofen on the postoperative analgesic requirements, pain intensity and other recovery parameters.

DETAILED DESCRIPTION:
The patients will be given general anaesthesia. Anaesthesia will be induced by propofol 1-2 mg/kg, and fentanyl 1-2 µg/kg. Endotracheal intubation will be facilitated by atracurium 0.5 mg/kg. Anaesthesia will be maintained by isoflurane in oxygen - air mixture. Transversus abdominis plane block will be performed at the end of the operation. A postoperative analgesic regimen according to group allocation will be started.

ELIGIBILITY:
Inclusion Criteria:

* American Society of anaesthesiologists physical status I to III.
* Open abdominal hysterectomy operations

Exclusion Criteria:

* History of gastrointestinal bleeding.
* History of intracranial haemorrhage.
* Pregnancy and lactation.
* Taking angiotensin converting enzyme(ACE) inhibitors or anticoagulation drugs.
* Asthmatic, hepatic,renal or heart failure.
* Abnormal platelet count.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2023-03-04 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Morphine consumption | Postoperative up to 24 hours
  mg

SECONDARY OUTCOMES:
Pain intensity | Postoperative up to 24 hours
  Visual analogue score: a score from 0 to 10( 0= no pain and 10 the worst imaginable pain)
Anaesthesia recovery time | Perioperative
  Minutes
Duration of post anaesthesia care unit stay | First postoperative 24 hours
  Minutes
Time of first ambulation | First postoperative 24 hours
  Minutes
Duration of hospital stay | Postoperative up to 4 weeks
  Days
Heart rate | Perioperative
  Beats/minute
Mean arterial blood pressure | Perioperative
  mmHg
Arterial oxygen saturation | Perioperative
  Percentage
End tidal carbon dioxide | Perioperative
  mmHg
Respiratory rate | Perioperative
  Breath/minute

CONTACTS AND LOCATIONS:
Overall Officials: Abd-Elazeem A Elbakry, MD, Principal Investigator — Menoufia University; Amal G Safan, MD, Principal Investigator — Menoufia University; Sadik A Sadik, MD, Principal Investigator — Menoufia University
Locations (1):
- Faculty of Medicine, Cairo, Shebin Elkom, Egypt